CLINICAL TRIAL: NCT01968395
Title: Pharmacokinetics of Caspofungin After One Dose in Patients With Liver Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E2013_PK_CASPO70_LIVERFAILURE
Record Dates: First submitted 2013-09-25; First posted 2013-10-24 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-06

CONDITIONS: Bacterial Infections and Mycoses; Liver Disease
MeSH Terms: conditions — Bacterial Infections and Mycoses; Liver Diseases | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Caspofungin 70 mg (Other): Infusion of one dose of Caspofungin 70 mg
  Interventions: Drug: Caspofungin 70 mg

INTERVENTIONS:
Drug: Caspofungin 70 mg — Intravenous use
  Other Names: Cancidas

SUMMARY:
The objective of this study is to conduct a population pharmacokinetic analysis of caspofungin in a population of patients with moderate and severe acute alcoholic hepatitis or liver disease with Child-Pugh score B and C in order to better characterize pharmacokinetic parameters in case of moderate and severe liver dysfunction.

DETAILED DESCRIPTION:
patients admitted for alcoholic hepatitis or decompensated cirrhosis and Child-Pugh score 7-9 and 10-15 will be included; all patients without invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Liver failure Child-Pugh B and C

Exclusion Criteria:

* Cachexia (BMI < 15 kg/m²)
* Pregnancy
* HIV
* Hepatitis C patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-10-21 (Actual)

PRIMARY OUTCOMES:
Measurement of serum caspofungine concentrations to determine the pharmacokinetic parameters of Caspofungin in patients with liver failure | 14 days
  one dose of caspofungin will be given to patients with hepatic failure. Serum sampling will be performed during 96 hours. Measurements of caspofungin in the serum will be performed to study the pharmacokinetics of this drugs and will be compared with pharmacokinetics of subjects with normal liver function. For safety, patients will be followed during 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique JACOBS, MD,PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium

REFERENCES:
- [Result] Gustot T, Ter Heine R, Brauns E, Cotton F, Jacobs F, Bruggemann RJ. Caspofungin dosage adjustments are not required for patients with Child-Pugh B or C cirrhosis. J Antimicrob Chemother. 2018 Sep 1;73(9):2493-2496. doi: 10.1093/jac/dky189. PMID 29860319